CLINICAL TRIAL: NCT04854265
Title: Effect of Mindfulness Meditation on Blood Pressure Among Young Hypertensive Adults
Brief Title: Mindfulness Meditation & Blood Pressure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universiti Tunku Abdul Rahman (Other)
Responsible Party: Principal Investigator, Imtiyaz Ali Mir, Principal Investigator, Universiti Tunku Abdul Rahman
Other Study IDs: U/SERC/171
Record Dates: First submitted 2021-04-13; First posted 2021-04-22 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Mindfulness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Mindfulness Meditation — Mindfulness meditation will include mindfulness based stress reduction program, Qigong, Tai Chi exercise, Yoga, and Pranayama breathing exercise.

SUMMARY:
Hypertension (HTN) is a common cardiovascular disorder present globally. In spite of various treatment approaches utilized in treating HTN, there is a surge in popularity of mindfulness meditation (MM) in recent years. Although multiple techniques of MM are advocated to be efficient in the treatment of HTN among hypertensive adults, the level of supportive evidence is variable and limited. Therefore authors aim to conduct a systematic review to investigate the effectiveness of mindfulness meditation on blood pressure (BP) among young adults.

DETAILED DESCRIPTION:
Hypertension (HTN) is one of the major culprit of cardiovascular disease and is potentially leading to premature death and disability globally, exerting tremendous burden to public health. A study in 2019 reported that globally, HTN affects 26% of world's population (972 million people), and the prevalence is expected to increase to approximately 29% by 2025, which is driven largely by increase in economically developing nations. World Health Organization (WHO) in year 2015 stated that there is 1 in every 4 men and 1 in every 5 women who had hypertension. A high prevalence of HTN highly cognate with diverse risk factors such as age, gender, ethnicity as well as other modifiable factors like unhealthy diet and physical inactivity.

Treatment of hypertension ranges from pharmacological approach to lifestyle changes. Antihypertensive medicines like Beta blockers, Calcium channel blocker, Alpha blockers, diuretics and angiotensin receptor blocker are casually used in controlling and lowering the blood pressure (BP). The cost of these ,medications is huge and are accompanied by many side effects. Due to this, HTN centered lifestyle modifications has now become a cornerstone as primary non-pharmacological first line therapy in the treatment of hypertension. Lifestyle modifications on HTN emphasize on smoking cessation, a healthy diet with more fruits and vegetables consumption, regular exercise of 10-20 minutes daily and so on. One of the lifestyle modification found to be effective and potentially able to reduce the high BP as potent as an antihypertensive drug is mindfulness meditation (MM). It is reported to reduce the diastolic BP by 2 mmHg which can significantly reduce the pervasiveness of HTN of about 17%, risk of befalling stroke by 15% and coronary heart disease by 6%.

There is no extensive peer-reviewed studies available to fortify the evidence of MM on HTN, as BP is affected by a combination of genetic, behavioral and environmental factors which cannot be easily controlled by meditation alone. In addition to that, to our knowledge no systematic reviews have been published on topic of MT effect on BP among hypertensive adults. Due to this, it is indispensable this study to be conducted to investigate the effect of MT in controlling BP among hypertensive adults.

This systematic review will adherence to Cochrane guidelines. We will conduct an extensive search of electronic databases such as the National Library of Medicine, Hindawi, Cochrane library, Cochrane library Central Register of Control Trial, MEDLINE, Pub Med and PEDro for eligible studies between 2000 to 2020. We will ensure that at least two bibliographic databases are involved for systematic review to avoid publication bias and promote generalizability of the results. To Attain optimal sensitivity and identify, all possible trials of MM on HTN, cluster of search terms will be created for the types of intervention (mindfulness or mindfulness meditations or Yoga or Tai Chi or QiGong) and another for population (Hypertension or high blood pressure). The clusters will be combined with AND and OR terms within the cluster.

In this systematic review, criteria for inclusion will be studies which are of randomized control trial design irrespective of type of MM used, any relevant studies published between year 2000 and 2020. In the aspect of sample population, adults whose age is between 18-60 years or mean age below 60 years will be selected. According to America Heart Association, only adults with stage 1 HTN (130-139/80-89 mmHg), stage 2 HTN (>140/90 mmHg) or HTN crisis (>180/120) will be chosen in this review regardless of the severity or type of HTN (primary or secondary). In addition, hypertensive patients with any other underlying health conditions (heart disease, chronic kidney disease) will be included in this study. Exclusion criteria will be studies published before 2000, studies which are not reported in English, studies which did not report BP as outcome measure, as well as BP measurement not implemented in a pre-test and post-test basis, studies which only report as abstract.

Qualitative analysis of the included studies will be used to establish narrative synthesis. Besides, we will also incorporate tabulation with narrative synthesis to allow comparison of findings to be made more easily. Post intervention differences in SBP and DBP between control and experimental group will be scrutinized descriptively by using measures of treatment effect.

ELIGIBILITY:
Inclusion Criteria:

- Adults aged 18-60 years with hypertension

Exclusion Criteria:

* Studies published before year 2000
* Not in English language
* Studies only reported with abstract

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Hypertensive adults (18-60years) who had undergone any kind of mindfulness meditation.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-05-04 (Actual); Primary Completion 2021-11-06 (Estimated); Study Completion 2021-12-24 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure | Change from Baseline Systolic Blood Pressure at 6 to 12 weeks
  Systolic blood taken from all the selected studies will be analyzed.
Diastolic blood pressure | Change from Baseline Diastolic Blood Pressure at 6 to 12 weeks
  Diastolic blood taken from all the selected studies will be analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Tunku Abdul Rahman, Kajang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ponte Marquez PH, Feliu-Soler A, Sole-Villa MJ, Matas-Pericas L, Filella-Agullo D, Ruiz-Herrerias M, Soler-Ribaudi J, Roca-Cusachs Coll A, Arroyo-Diaz JA. Benefits of mindfulness meditation in reducing blood pressure and stress in patients with arterial hypertension. J Hum Hypertens. 2019 Mar;33(3):237-247. doi: 10.1038/s41371-018-0130-6. Epub 2018 Nov 13. PMID 30425326
- See also: Hypertension Prevalence — https://www.who.int/news-room/fact-sheets/detail/hypertension